CLINICAL TRIAL: NCT02663102
Title: Assessment of Safety of GlaxoSmithKline (GSK) Vaccines' Quadrivalent Seasonal Influenza Vaccine, Fluarix Tetra When Administered According to the Approved Prescribing Information in Korea.
Brief Title: Evaluation of Safety of GlaxoSmithKline (GSK) Vaccines' Quadrivalent Seasonal Influenza Vaccine, Fluarix Tetra When Administered According to the Approved Prescribing Information (PI) in Korea.
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 204687
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-10

CONDITIONS: Influenza, Human
Keywords: Safety; Post-marketing; Korea; Drug utilization study; Fluarix Tetra
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Fluarix Tetra Group 1: Subjects aged between 6-35 months old who received Fluarix Tetra as per locally approved PI (which is not part of the drug use investigation).
  Interventions: Other: Data collection
- Fluarix Tetra Group 2: Subjects aged 3 years and above who received Fluarix Tetra as per locally approved PI (which is not part of the drug use investigation).
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Safety monitoring and evaluation: - Recording of all AEs during the study period using diary cards, follow-up contact via telephone or email. - Recording of SAEs throughout the study period for each subject.

SUMMARY:
The purpose of this study is to collect safety information on the use of Fluarix Tetra according to the approved PI, in Korea, over a period of 6 years from children greater than or equal to (≥)3 years of age and adults, and over a period of 4 years from children between 6 months and 35 months of age.

DETAILED DESCRIPTION:
Adults and previously vaccinated children aged ≥6 months, a single dose of Fluarix Tetra will be administered. To previously unvaccinated children aged 6 months to less than (<) 9 years, two doses will be administered with a second dose at least 4 weeks apart from the first one as per the local PI in Korea.

Fluarix Tetra may be administered to pregnant women/lactating women as per PI, if there is a clear need. Pregnancy outcome (whether full-term or premature, information on the status of the mother and child) in vaccinated pregnant subjects will be followed-up at 6-8 weeks after delivery, if possible.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who were vaccinated with Fluarix Tetra or eligible to receive Fluarix Tetra according to the locally approved PI.
* Signed informed consent as Informed Consent Form (ICF)/Informed Assent Form (IAF) obtained from the subject/subject's parent(s)/Legally acceptable Representative(s) [LAR(s)].

Exclusion Criteria:

* Those who are not eligible for vaccination with Fluarix Tetra according to the local PI.

  * Hypersensitivity reaction to Fluarix Tetra.
  * History of hypersensitivity reaction to Influenza vaccine.
  * History of Guillain-Barre syndrome or other nervous system abnormalities to Influenza vaccine within 6 weeks post-vaccination.
* Those who are not eligible for vaccination with Fluarix Tetra according to the medical judgement of physician.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy subjects aged 6 months and above who were vaccinated with Fluarix Tetra or eligible to receive Fluarix Tetra in Korea according to the locally approved PI.
Sampling Method: Non-Probability Sample
Enrollment: 1388 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- South Korea (10):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Donghae
  - GSK Investigational Site, Gwangmyeong
  - GSK Investigational Site, Gyeongsangbuk-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon-si, Gyeonggi-do
  - GSK Investigational Site, Ulsan
  - GSK Investigational Site, Yangju-si, Gyeonggi-do

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluarix Tetra Group 1 | Fluarix Tetra Group 2
Started | 687 | 701
Completed | 687 | 701
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix Tetra Group 1 | Fluarix Tetra Group 2 | Total
Number analyzed (Participants) | 687 | 701 | 1388
Age, Customized [Count of Participants; unit: Participants]
  6 months - 11 months | 275 | 0 | 275
  >1 year - <2 years | 233 | 0 | 233
  >2 years - < 3 years | 179 | 0 | 179
  3 years - 9 years | 0 | 167 | 167
  10 years - 19 years | 0 | 89 | 89
  20 years - 29 years | 0 | 56 | 56
  30 years - 39 years | 0 | 108 | 108
  40 years - 49 years | 0 | 104 | 104
  50 years or more | 0 | 177 | 177
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 323 | 376 | 699
  Male | 364 | 325 | 689
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 686 | 701 | 1387
  Non-Korean | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Expected Adverse Events (AEs)
Description: An adverse event that is expected from the subject during the post-vaccination follow-up period as described in the locally approved Prescribing Information.
Time Frame: During the 21 days follow-up period after vaccination (i.e. day of vaccination and 20 subsequent days)
Population: The analysis was performed on the Safety analysis set which included all subjects who received Fluarix Tetra, participated in the drug use investigation and provided post vaccination safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Tetra Group 1 | Fluarix Tetra Group 2
Number analyzed (Participants) | 687 | 701
Participants | 54 | 44

2. Primary Outcome: Number of Participants With Unexpected Adverse Events (AEs)
Description: Any adverse event reported in addition to those expected during the drug use investigation. Adverse events that are not reflected in the approved Prescribing Information.
Time Frame: During the 21 days follow-up period after vaccination (i.e. day of vaccination and 20 subsequent days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Tetra Group 1 | Fluarix Tetra Group 2
Number analyzed (Participants) | 687 | 701
Participants | 116 | 62

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAEs assessed included any adverse event that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the 21 days follow-up period after vaccination (i.e. day of vaccination and 20 subsequent days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Tetra Group 1 | Fluarix Tetra Group 2
Number analyzed (Participants) | 687 | 701
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Solicited and Unsolicited AEs were collected during the 21-day follow-up period after each vaccination. SAEs were collected from the date of vaccination in the drug use investigation up to 21 days (Day 0 to Day 20) after vaccination of the subject in the drug use investigation.
Arm/Group | Fluarix Tetra Group 1 | Fluarix Tetra Group 2
All-Cause Mortality (participants affected / at risk) | 0/687 | 0/701
Serious Adverse Events (participants affected / at risk) | 3/687 | 1/701
Other Adverse Events (participants affected / at risk) | 167/687 | 105/701
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluarix Tetra Group 1 (N=687) | Fluarix Tetra Group 2 (N=701)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Kawasaki's disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluarix Tetra Group 1 (N=687) | Fluarix Tetra Group 2 (N=701)
Nasopharyngitis (Infections and infestations) | 49 (53) | 17 (17)
Rhinitis (Infections and infestations) | 23 (23) | 4 (4)
Bronchitis (Infections and infestations) | 19 (19) | 9 (9)
Acute sinusitis (Infections and infestations) | 5 (5) | 0 (0)
Otitis media acute (Infections and infestations) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3)
Bronchiolitis (Infections and infestations) | 3 (3) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (3) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 5 (5)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 5 (5)
Myringitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 3 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (3)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 7 (7) | 9 (9)
Pyrexia (General disorders) | 33 (35) | 8 (8)
Administration site pruritus (General disorders) | 2 (2) | 3 (3)
Injection site erythema (General disorders) | 2 (2) | 3 (3)
Administration site induration (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 9 (9)
Injection site warmth (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1)
Enteritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spams (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 3 (3) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT02663102/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT02663102/SAP_001.pdf